CLINICAL TRIAL: NCT02955589
Title: A Phase 2b Open-Label Single-Arm Study to Evaluate the Efficacy and Safety of Oral HBI-8000 in Patients With Relapsed or Refractory Adult T Cell Lymphoma (ATL)
Brief Title: Efficacy and Safety of Oral HBI-8000 in Patients With Relapsed or Refractory Adult T Cell Lymphoma (ATL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HUYABIO International, LLC. (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBI-8000-210
Record Dates: First submitted 2016-11-01; First posted 2016-11-04 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Adult T-Cell Lymphoma (ATL)
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — HBI-8000

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HBI-8000 (Experimental): Four 10 mg tablets or less twice weekly orally approximately 30 minutes after any regular meal. The treatment will be continuous, with 3-4 days between dosing. Treatment will continue until disease progression in the absence of unacceptable toxicity.
  Interventions: Drug: HBI-8000

INTERVENTIONS:
Drug: HBI-8000 — Oral, twice weekly

SUMMARY:
Phase 2b, open-label, non-randomized, single arm study to evaluate the safety, and efficacy of HBI-8000 40 mg BIW in patients with relapsed or refractory ATL (R/R ATL)

DETAILED DESCRIPTION:
This is a Phase 2b, open-label, non-randomized, single arm study to evaluate the safety, and efficacy of HBI-8000 40 mg BIW in patients with relapsed or refractory ATL (R/R ATL). HBI 8000 will be administered orally approximately 30 minutes after any regular meal twice a week. There will be 3 to 4 days between dosing. A treatment cycle is defined as 28 consecutive days. HBI-8000 administration will be continued until disease progression or unacceptable toxicities are observed despite appropriate dose reduction or treatment interruption.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathological, or cytological diagnosis of ATL confirmed as seropositive for anti-Human T-lymphotrophic Virus type-I (HTLV-I) antibody
2. Acute, lymphoma or unfavorable chronic types. The unfavorable chronic type is defined by the presence of at least 1 of the following: serum albumin <3.5 g/dL, lactic dehydrogenase (LDH) >300 U/L, or blood urea nitrogen (BUN) >25 mg/dL. The patient must have at least 1 of measurable lesion, or evaluable lesion in either of peripheral blood or skin
3. Relapsed or refractory disease after receiving prior systemic therapy with mogamulizumab, or ≥1 prior systemic therapy with cytotoxic chemotherapy in case of intolerance/contraindication for mogamulizumab. And there is no other standard treatment which can be considered appropriate for patients
4. Male or female, aged 20 years or older
5. ECOG Performance Status of 0-2
6. Life expectancy of greater than 3 months
7. Meeting the following baseline laboratory criteria for screening:

   * Absolute Neutrophil Count >1500/µL independent of growth factor support within 7 days
   * Platelets >75,000/µL independent of transfusion within 14 days
   * Hgb >8 g/dL independent of transfusion within 14 days
   * Serum creatinine < 1.5 X upper limit of normal (ULN)
   * Serum aspartate aminotransferase/glutamyl oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase/glutamyl pyruvic transaminase (ALT/SGPT) less than or equal to 3 X ULN
   * Serum Bilirubin less than or equal to 1.5 X ULN
8. Negative serum pregnancy test for females of childbearing (reproductive) potential. Female patients of child bearing potential must use an effective method of birth control (e.g., hormonal contraceptive, intrauterine device, diaphragm with spermicide or condom with spermicide) during treatment period and 1 month thereafter; Males must use an effective method of birth control (2 barrier methods) during treatment period and 3 months thereafter.

   Note: Female patients will be considered to be women of childbearing potential unless having undergone permanent contraception or postmenopausal. Postmenopausal is defined as at least 12 months without menses with no other medical reasons (e.g., chemical menopause because of treatment with anti-malignant tumor agents).
9. Signed informed consent

Exclusion Criteria:

2.5.2 Exclusion Criteria:

1. Patients in whom central nervous system lymphoma is recognized during screening (if suspected clinically, imaging study should be performed to confirm)
2. Male patients with QTcF > 450 msec at screening, female patients with QTcF > 470 msec at screening, or patients with congenital long QT syndrome, clinically significant arrhythmia, history of congestive heart failure (New York Heart Association Class III or IV) or acute myocardial infarction within 6 months of starting the study drug at screening.
3. Patients with known hypersensitivity to benzamide class of compounds or any of the components of HBI-8000 tablets, and patients with prior exposure of HBI-8000;
4. Patients with a history of second malignancy other than disease under study. The exceptions are disease (excluding disease listed below) that has been treated with curative intent with no evidence of recurrence in past 5 years. Furthermore, if the second malignancy is one of the following diseases that were treated with curative intent, it is only required that there is no evidence of recurrence in past 2 years;

   * Basal cell carcinoma of the skin
   * Squamous cell carcinoma of the skin
   * Cervical carcinoma in situ
   * Carcinoma in situ of the breast
   * An incidental histological finding of prostate carcinoma (TNM stage T1a or T1b)
   * Early-stage gastric cancer treated with endoscopic mucosal resection or endoscopic submucosal dissection
5. Autologous stem cell transplantation within 12 weeks (84 days) of starting the study drug
6. History of allogeneic stem cell transplantation
7. Organ transplantation recipients except autologous hematopoietic stem cell transplantation
8. Uncontrolled inter-current infection
9. Hepatitis B surface antigen-positive, or hepatitis C virus antibody positive. In case hepatitis B core antibody and/or hepatitis B surface antibody is positive even if hepatitis B surface antigen negative, a hepatitis B virus DNA test (real-time PCR measurement) should be performed and if positive, the patient should be excluded from study
10. Any history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
11. Uncontrolled diabetes mellitus, hypertension, endocrine disorder, bleeding disorder
12. Major surgery or radiation therapy within 28 days of starting the study drug
13. Receiving investigational agents or anti-cancer therapy within 28 days, nitrosourea or mitomycin C within 42 days, of starting the study drug
14. Receiving antibody therapy for ATL within 4 weeks of starting the study drug
15. Women who are breastfeeding or women who are not willing to stop breastfeeding during study treatment period and for 30 days after the last dose of study drug
16. Potential for non-compliance or at increased risk based on investigator's judgement

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-11; Primary Completion 2018-12 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Lee, MD, Study Chair — HUYA Bioscience International, LLC
Locations (15):
- Japan (15):
  - Fukuoka
  - Isehara
  - Kagoshima
  - Miyagi
  - Miyazaki
  - Nagasaki
  - Nagoya
  - Okinawa
  - Ōita
  - Ōmura
  - Saitama
  - Sapporo
  - Suita
  - Tokyo
  - Yufu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Utsunomiya A, Izutsu K, Jo T, Yoshida S, Tsukasaki K, Ando K, Choi I, Imaizumi Y, Kato K, Kurosawa M, Kusumoto S, Miyagi T, Ohtsuka E, Sasaki O, Shibayama H, Shimoda K, Takamatsu Y, Takano K, Yonekura K, Makita S, Taguchi J, Gillings M, Onogi H, Tobinai K. Oral histone deacetylase inhibitor tucidinostat (HBI-8000) in patients with relapsed or refractory adult T-cell leukemia/lymphoma: Phase IIb results. Cancer Sci. 2022 Aug;113(8):2778-2787. doi: 10.1111/cas.15431. Epub 2022 Jun 7. PMID 35579212

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One more patient than planned consented.
Period: Overall Study
Arm/Group | HBI-8000
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Arm/Group | HBI-8000
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.4 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 23
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 23
Sub-Type of ATL at Screening [Count of Participants; unit: Participants]
  Acute ATL | 13
  Lymphoma ATL | 8
  Unfavorable Chronic ATL | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response rate (CR+CRu+PR) was determined based on the response of all compartments (lymph nodes, extranodal masses, spleen & liver, skin, peripheral blood, and bone marrow) per Tsukasaki criteria and skin lesions were evaluated according to modified SWAT.
  CR: The disappearance of all disease whereby all criteria met; All compartments are normal.
  CRu: Lymph nodes ≥75% decrease and extranodal masses ≥75% decrease, but presence of residual lesion; spleen, liver, skin, peripheral blood and bone marrow are normal.
  PR: Lymph nodes and extradnodal masses - Reduction rate of the sum of 2 dimension products of ≥50% and ≤75%, no increase spleen /liver, skin lesion ≥50% decrease and peripheral blood ≥50% decrease.
Time Frame: Tumor response was assessed until disease progression or unacceptable toxicity, up to 15 months.
Population: Per Protocol Set
Measure: Count of Participants; unit: Participants
Arm/Group | HBI-8000
Number analyzed (Participants) | 23
Participants | 7

2. Secondary Outcome: Objective Response Rate by Disease Subtype
Description: Objective response rate (CR+CRu+PR) by disease subtype (acute ATL, lymphoma ATL, unfavorable chronic ATL) was determined based on the response of all compartments (lymph nodes, extranodal masses, spleen & liver, skin, peripheral blood, and bone marrow) per Tsukasaki criteria and skin lesions were evaluated according to modified SWAT.
Time Frame: Tumor response was assessed until disease progression or unacceptable toxicity, up to 15 months.
Population: Per Protocol Set
Measure: Count of Participants; unit: Participants
Groups:
- HBI-8000 Acute ATL; HBI-8000 Lymphoma ATL; HBI-8000 Unfavorable Chronic ATL: Four 10 mg tablets or less twice weekly orally approximately 30 minutes after any regular meal. The treatment will be continuous, with 3-4 days between dosing. Treatment will continue until disease progression in the absence of unacceptable toxicity.
  HBI-8000: Oral, twice weekly
Arm/Group | HBI-8000 Acute ATL | HBI-8000 Lymphoma ATL | HBI-8000 Unfavorable Chronic ATL
Number analyzed (Participants) | 13 | 8 | 2
Participants | 6 | 1 | 0

3. Secondary Outcome: Median Duration of Progression-free Survival (PFS)
Description: PFS was defined as the duration from the date of the first study drug dose to the disease progression or death, whichever occurs first. Evaluation of progression/progressive disease is performed according to the modified criteria of the International Consensus Meeting. Progression is defined as a 50% increase in the sum of 2-dimension products of nodal and/or extra nodal lesions, or 25% increase of mSWAT score in skin lesion, or 50% increase of absolute count of abnormal lymphocyte, or the appearance of new lesions.
Time Frame: From the first day of HBI-8000 dose to the day of disease progression or death, which ever came first, through the end of the study (up to 15 months).
Population: Per Protocol Set
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | HBI-8000
Number analyzed (Participants) | 23
Weeks | 7.6 [3.4 to 32.1]

4. Secondary Outcome: Median Duration of Response (DOR)
Description: Median duration of response from first response CR, CRu, PR, date to progression, death or last available tumor assessment.
Time Frame: Through the end of the study (up to 12 months).
Population: Per Protocol Set
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | HBI-8000
Number analyzed (Participants) | 23
Weeks | 40.0 [11.4 to NA] — Upper limit was not reached due to insufficient number of participants with events

5. Other Pre Specified Outcome: Median Duration of Overall Survival (OS)
Description: Median duration of overall survival is from start of the study to death.
Time Frame: Until death, assessed every 3 months up to 12 months after last treatment through the end of the study (up to 30 months).
Population: Per Protocol Set
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | HBI-8000
Number analyzed (Participants) | 23
Weeks | 34.4 [10.1 to 78.3]

6. Other Pre Specified Outcome: Safety and Tolerability, Evaluated as Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Safety and tolerability, evaluated as number of participants with treatment-related adverse events as assessed by CTCAE v4.0.
Time Frame: From date of first subject's consent until 30 days after last treatment, assessed up to 25 months.
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | HBI-8000
Number analyzed (Participants) | 23
Participants | 23

ADVERSE EVENTS:
Time Frame: From date of the first subject's consent to 12 months after last treatment, assessed up to 36 months.
Arm/Group | HBI-8000
All-Cause Mortality (participants affected / at risk) | 16/23
Serious Adverse Events (participants affected / at risk) | 7/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HBI-8000 (N=23)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HBI-8000 (N=23)
Anaemia (Blood and lymphatic system disorders) | 8 (19)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (29)
Diarrhoea (Gastrointestinal disorders) | 6 (7)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (4)
Malaise (General disorders) | 7 (10)
Pyrexia (General disorders) | 3 (5)
Fatigue (General disorders) | 3 (6)
Platelet count decreased (Investigations) | 15 (64)
Neutrophil count decreased (Investigations) | 11 (53)
White blood cell count decreased (Investigations) | 9 (47)
Weight decreased (Investigations) | 4 (6)
Aspartate aminotransferase increased (Investigations) | 2 (3)
Gamma-glutamyltransferase increased (Investigations) | 2 (5)
Lymphocyte count decreased (Investigations) | 2 (11)
Decreased appetite (Metabolism and nutrition disorders) | 8 (11)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Huya has agreements with PIs and the agreements restricts the right of the PI to discuss or publish trial results after the trial is completed.

The content of disclosure restriction stated in the agreement is "PI shall obtain sponsor's prior written consent before disclosing the information obtained from this clinical trial to a professional society or other external party."

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT02955589/Prot_SAP_000.pdf